CLINICAL TRIAL: NCT07185958
Title: Dual Energy CT - a Tool for Delineation of Tumor and Organs at Risk in Radiotherapy
Acronym: DART
Status: Not yet recruiting | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Collaborators: Copenhagen University Hospital at Herlev (Other); Odense University Hospital (Other)
Responsible Party: Principal Investigator, Hella Maria Brøgger Sand, Principal Investigator, Aalborg University Hospital
Other Study IDs: N-20250004
Record Dates: First submitted 2025-09-07; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Brain Metastases; Bone Metastases; Head and Neck Cancer; Lung Cancer
Keywords: tumor delineation; organs at risk delineation; dual-energy CT; DECT; radiotherapy
MeSH Terms: conditions — Brain Neoplasms; Head and Neck Neoplasms; Lung Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- DART Brain (whole): Patients with 1-5 brain metastases referred for whole brain radiotherapy. Intervention: Extra DECT scan with iodine-based contrast agent + extra MRI scan with Gadolinium-based contrast agent.
  Interventions: Diagnostic Test: Dual-energy CT (DECT); Drug: Iodine-based contrast agent; Diagnostic Test: Magnetic Resonance Imaging (MRI); Drug: Gadolinium-based contrast agent
- DART Brain (SRS): Patients with 1-5 brain metastases referred for stereotactic radiotherapy. Intervention: Extra DECT scan with iodine-based contrast agent.
  Interventions: Diagnostic Test: Dual-energy CT (DECT); Drug: Iodine-based contrast agent
- DART Bone (pall): Patients with bone metastases without medullary involvement in one or more regions of the vertebral column (C1-C7, Th1-12, L1-L5, Os Sacrum) referred for palliative radiotherapy. Intervention: Extra DECT scan with iodine-based contrast agent + extra MRI scan without contrast agent.
  Interventions: Diagnostic Test: Dual-energy CT (DECT); Drug: Iodine-based contrast agent; Diagnostic Test: Magnetic Resonance Imaging (MRI)
- DART Bone (SBRT): Patients with bone metastases without medullary involvement in one or more regions of the vertebral column (C1-C7, Th1-12, L1-L5, Os Sacrum) referred for palliative radiotherapy. Intervention: Extra DECT scan with iodine-based contrast agent.
  Interventions: Diagnostic Test: Dual-energy CT (DECT); Drug: Iodine-based contrast agent
- DART H&N: Patients with head and neck cancer referred for radiotherapy. Patients must have undergone a PET/CT scan during the diagnostic evaluation for cancer. Intervention: Extra DECT scan without contrast agent.
  Interventions: Diagnostic Test: Dual-energy CT (DECT)
- DART Lung: Patients with lung cancer referred for palliative radiotherapy with a maximum of 10 fractions. Interventions: Extra DECT scan in breath-hold without contrast agent.
  Interventions: Diagnostic Test: Dual-energy CT (DECT)

INTERVENTIONS:
Diagnostic Test: Dual-energy CT (DECT) — Additional DECT scan performed for tumor and OAR delineation.
Drug: Iodine-based contrast agent — Administered intravenously with DECT for enhanced imaging.
  Groups: DART Bone (SBRT); DART Bone (pall); DART Brain (SRS); DART Brain (whole)
Diagnostic Test: Magnetic Resonance Imaging (MRI) — Additional MRI scan performed for tumor and OAR delineation.
  Groups: DART Bone (pall); DART Brain (whole)
Drug: Gadolinium-based contrast agent — Administered intravenously with MRI for enhanced imaging.
  Groups: DART Brain (whole)

SUMMARY:
The primary aim of this clinical study, 'Dual Energy CT - a tool for delineation of tumor and organs at risk in radiotherapy' (DART) is to evaluate whether dual-energy CT (DECT) is at least as effective as magnetic resonance imaging (MRI) in delineating both tumors and organs at risk (OARs) in patients referred for radiotherapy (RT). This primary aim will be explored in patient groups where the performance of DECT for RT has been described in the literature (but mostly based on signal-to-noise ratio and/or contrast-to-noise ratio), such as brain metastases (sub-cohort 'DART Brain') and head and neck cancer (sub-cohort 'DART H&N'). Additionally, DART will explore diagnoses not yet studied in the literature, such as bone metastases (sub-cohort 'DART Bone'). If DECT could be demonstrated to achieve delineations for RT in both tumors and OARs that are equally accurate as those based on MRI, it could offer significant advantages by being faster and more cost-effective, making DECT a valuable alternative to MRI in clinical practice. As a secondary aim, the study will evaluate whether DART offers benefits when added to standard RT imaging for tumor and OAR delineation: (1) For lung cancer patients (sub-cohort 'DART Lung'), where MRI scans are typically not valuable due to tumor motion caused by breathing, 'DART Lung' will assess whether DECT performed in breath-hold provides added value compared to the single-energy CT (SECT) scan conducted during free breathing, as used in current clinical practice. (2) For head and neck cancer patients, 'DART H&N' will evaluate whether DECT offers added value compared to the positron emission tomography (PET)/CT scan currently used in clinical practice.

DETAILED DESCRIPTION:
A detailed description of the study is provided in the uploaded document 'Study Protocol with Statistical Analysis Plan'.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status (PS) 0-2
* Assessed to be able to complete the protocol scanning regime
* Referred for RT
* For head and neck cancer patients, a PET/CT scan must have been performed during the diagnostic evaluation for cancer
* Signed informed consent

Exclusion Criteria:

* Pregnancy
* Previous RT in the same anatomical area now referred for RT
* Previous surgery in the same anatomical area now referred for RT
* Participation in conflicting protocols
* If relevant for the protocol scanning regime: Allergic to contrast agent
* If relevant for the protocol scanning regime: Contraindication to iodine-based contrast agent for CT (as determined by the physician)
* If relevant for the protocol scanning regime: Contraindication to Gadolinium-based contrast agent for MRI (as determined by the physician)
* If relevant for the protocol scanning regime: Contraindication for MRI (pacemaker, metal, non-MRI, compatible implants etc.)
* Incapable of understanding the patient information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients referred for radiotherapy at Aalborg University Hospital, Denmark. For the 'DART Bone (SBRT)' cohort, patients are also referred for radiotherapy at Odense University Hospital and Copenhagen University Hospital, Herlev and Gentofte, Denmark
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-09-22 (Estimated); Primary Completion 2028-03-21 (Estimated); Study Completion 2028-03-21 (Estimated)

PRIMARY OUTCOMES:
Inter-observer variability (geometric differences in volume and surface) of manual tumor and OAR delineations on DECT compared with SECT/MRI. | Baseline (time of imaging before radiotherapy planning)
  For patients enrolled in cohorts 'DART Brain', 'DART Bone' and 'DART H&N', the accuracy of manual delineations of tumors and OARs on DECT scans will be compared to those manually performed on a combination of SECT and MRI scans for each patient. For patients enrolled in 'DART H&N' the comparison will also be done to the PET/CT scan.
  A reduction in inter-observer variability in delineations will serve as an indicator of improved contour accuracy for both tumors and OARs. Inter-observer variability for tumor and OAR delineations on DECT and SECT/MRI scans, respectively, will be measured as geometric differences between individual manual delineations and consensus structures for each tumor and OAR. Consensus structures will be generated on both DECT and SECT/MRI scans using the STAPLE function with a 50% agreement threshold. Variations relative to the consensus structures will be reported using various metrics, including volume and surface differences.

SECONDARY OUTCOMES:
Qualitative image-quality assessment of tumors and OARs using a Likert scale (or comparable method) for DECT compared with SECT/MRI. | Baseline (time of imaging before radiotherapy planning)
  The secondary outcome will be measured in all patient cohorts ('DART Brain', 'DART Bone', 'DART H&N', and 'DART Lung'). Image-quality for tumors and OARs will be evaluated qualitatively by experienced oncologists using a Likert scale or comparable method, and evaluations will be made and reported between DECT and SECT/MRI scans (and, for patients enrolled in 'DART H&N', also PET/CT scans).

CONTACTS AND LOCATIONS:
Overall Officials: Hella MB Sand, Medical Physicist, MSc, Principal Investigator — Department of Medical Physics, Oncology, Aalborg University Hospital, Aalborg, Denmark
Locations (3):
- Denmark (3):
  - Aalborg University Hospital, Aalborg
  - Copenhagen University Hospital Herlev and Gentofte, Herlev
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-30): https://cdn.clinicaltrials.gov/large-docs/58/NCT07185958/Prot_SAP_000.pdf